CLINICAL TRIAL: NCT06835114
Title: Different Surgical Strategies for Management of Severely Diseased Left Anterior Descending Artery During Coronary Artery Bypasses Grafting
Brief Title: Reconstruction of Diffusely Diseased Left Anterior Descending with Left Internal Mammary Artery On-lay Patch or Saphenous Vein Patch Without Endarterectomy by Opening the Whole Wall of the Diseased Segment(s) Has Less Risk and Fewer Complications Compared to Endarterectomy Technique
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Ibrahim Gadallah, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Left anterior descending
Record Dates: First submitted 2024-12-09; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: LAD (Left Anterior Descending) Coronary Artery Stenosis
MeSH Terms: conditions — Leukocyte adhesion deficiency type 1; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Management of severly diseased LAD (Experimental): Different surgical strategies for management of severly diseased LAD
  Interventions: Procedure: CABG; Procedure: LIMA on lay patch; Procedure: Safenous vein patch

INTERVENTIONS:
Procedure: CABG — CABG
Procedure: LIMA on lay patch — Left internal mammary artery harvesting with on lay patch on left anterior descending coronary artery
Procedure: Safenous vein patch — Safenous vein patch on left anterior descending artery

SUMMARY:
The objective of this study is to compare different surgical strategies for management of severely diseased LAD artery during CABG i.e. LIMA on-lay patch vs. saphenous vein patch and the distal in situ LIMA and saphenous vein graft (LIMA+ SVG).

DETAILED DESCRIPTION:
Total myocardial revascularization is the primary aim of coronary artery bypass grafting (CABG) . Conventional CABG does not attain sufficient myocardial revascularization in severely diseased left anterior descending coronary artery (LAD). Coronary endarterectomy for severely atherosclerotic LAD was first introduced by Bailey and his coworkers , but it has a higher risk of morality and poor outcomes. The reconstruction of LAD with saphenous vein or left internal mammary artery (LIMA) combined with endarterectomy was described by Fundaro and others surgeons for better long-term patency of LIMA graft and to avoid the drawbacks of endarterectomy. Reconstruction of diffusely diseased LAD with LIMA on-lay patch or saphenous vein patch without endarterectomy by opening the whole wall of the diseased segment(s) has less risk and fewer complications compared to endarterectomy technique. However, the superiority of LIMA path versus saphenous vein patch is still controversial.

In addition, the LIMA patch is occasionally not available as a bypass to LAD, for example with relatively shorter LIMA due to enlarged left ventricle, difficulty in harvesting the proximal LIMA, accidental injury of the LIMA pedicle during harvesting, calcification of the middle or distal LIMA or mismatching between the LAD and distal LIMA. To overcome this, an end-to-end anastomosis with the distal in situ LIMA and saphenous vein graft (SVG) was performed to establish a composite graft to bypass the LAD.

ELIGIBILITY:
Inclusion Criteria:

* included patients with long-segment diffusely diseased LAD, with good ejection fraction and elective surgery.

Exclusion Criteria:

* Patients with associated valve surgery, left ventricular EF less than 40%, and severe comorbidities (renal or liver failure), preoperative dialysis, and hemodynamic instability, emergency operations were excluded.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-12-10 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Serum troponin level | From enrollment to 1 month after intervention
  Measure serum troponin level after 48h , after 1 week and after 1 month